CLINICAL TRIAL: NCT00238680
Title: The Effect of Programmable Timer in Bladder Rehabilitation Treatment of Idiopathic Overactive Bladder in Children
Brief Title: Programmable Timer in the Bladder Rehabilitation Treatment of OAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHTIMER2005; 2005-41-4853, 20040192
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Overactive Bladder; Urinary Incontinence
Keywords: Overactive bladder; Children; Bladder rehabilitation
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence

INTERVENTIONS:
Behavioral: Bladder rehabilitation
Behavioral: Bladder rehabilitation with programmable timer

SUMMARY:
The purpose of this study is to evaluate the effect of bladder rehabilitation in a non-selected group of children with idiopathic overactive bladder and to clarify whether the effect of the treatment can be increased by addition of a programmable timer

DETAILED DESCRIPTION:
Daytime urinary incontinence is common in children. At the age of 7 a prevalence of 2-9 % has been reported. Daytime urinary incontinence is a heterogenic multifactorial illness where the the symptoms has several degrees of severity and can be caused by different mechanisms. Daytime urinary incontinence can be etiologically classified in the rare neurogenic and structural forms and the common functional or idiopathic form (where no neurological or structural cause of the bladder dysfunction can be identified.

The symptom based diagnosis OAB (overactive bladder) is most often used to describe daytime urinary incontinence in children. OAB is defined as a symptom syndrome including urgency with or without urge incontinence in combination with frequency.

When urinary tract infection and neurogenic and structural causes has been excluded the nonpharmacological bladder rehabilitation is first line treatment in children with OAB. It is expected that approximately 50 % of the children can be relieved of symptoms by this treatment. The treatment consist of instruction in good micturition habits including toilet position, sufficient fluid intake and voidings at predefined intervals. The treatment effect is to a large degree dependent upon the ability of the children to void at fixed intervals. Children at the age of 5-10 yrs generally find this difficult and a programmable timer seems be an useful instrument in order to remind the child of voiding at fixed times. However there has not been published studies of the effect of programmable timer.

Hypothesis:

* Daytime urinary incontinence in children aged 5-15 with idiophatic OAB can in 50 % of cases be cured by bladder rehabilitation
* The compliance of the bladder rehabilitation treatment can for each individual be increased by adding a programmable timer to the treatment.

Material and methods:

100 children with idiopathic OAB will be recruited from the Center of Child Incontinence, Skejby University Hospital, Aarhus, Denmark.

After a run-in period of at least 4 weeks the children will be randomized to 12 weeks of bladder rehabilitation with or without programmable timer.

The effect of the treatment will be estimated based on home recordings.

ELIGIBILITY:
Inclusion Criteria:

* Daytime urinary incontinence with at least 1 episode of at least 1 ml per week
* More than 6 voidings per day
* Informed consent

Exclusion Criteria:

* Known diseases of the kidneys or urinary tract besides OAB
* Receiving treatment with drugs that have an effect on the urine production or bladder function

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100
Dates: Start 2005-03; Primary Completion 2006-09 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Clinical effects evaluated by home registrations of incontinence episodes and frequency volume charts at specified intervals.

SECONDARY OUTCOMES:
Bladder capacity measure before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Soeren Hagstroem, MD, Principal Investigator — University of Aarhus
Locations (1):
- Department of pediatrics, University hospital of Aarhus, Skejby Sygehus, Aarhus, Aarhus N, Denmark